CLINICAL TRIAL: NCT05699226
Title: Amplitude Titration to Improve ECT Clinical Outcomes Randomized Clinical Trial
Brief Title: Amplitude Titration to Improve ECT Clinical Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R33MH125126 (NIH); 5R61MH125126 (NIH)
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Depression; ECT; Cognitive Change
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two arms: experimental (variable amplitude) and control (fixed amplitude). Participant and outcomes assessor will be masked to assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: This investigation will use allocation concealment and masking for subject assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Variable amplitude (Experimental): Individualized amplitude
  Interventions: Device: Soterix Medical Incorporated 4x1 adapter
- Fixed amplitude (Active Comparator): Fixed (800 milliamperes) amplitude
  Interventions: Device: Traditional ECT device

INTERVENTIONS:
Device: Soterix Medical Incorporated 4x1 adapter — Device permits individualized amplitudes
  Arms: Variable amplitude
Device: Traditional ECT device — FDA approved ECT device with fixed amplitude.
  Arms: Fixed amplitude

SUMMARY:
A randomized controlled trial will compare hippocampal neuroplasticity, antidepressant, and cognitive outcomes between individualized amplitude and fixed 800 mA amplitude ECT in older depressed subjects (n = 25 per group, n = 50 total). Relative to fixed 800 mA ECT:

H1: Individualized amplitude arm will have improved RUL antidepressant outcome (IDS-C30 response rates and reduced BT electrode placement switch at V2).

H2: Individualized amplitude arm will have improved cognitive outcomes (DKEFS-Verbal Fluency

DETAILED DESCRIPTION:
ECT dosing can be divided into three categories for the ECT responder: insufficient (no antidepressant response, no cognitive impairment), optimal (antidepressant response, no cognitive impairment), or excessive (antidepressant response, cognitive impairment). Traditional fixed amplitude ECT dosing with 800 mA adjusts pulse train duration and frequency based on seizure titration or demographic factors (age, sex). Fixed amplitude produces variable electric fields and ECT dosing secondary to individual neuroanatomic differences. Adjustments to pulse width, pulse train duration, and frequency do not improve the efficacy of insufficient dosing or mitigate the cognitive risk of excessive dosing. In contrast, individualized amplitude based on electric field modeling or amplitude seizure titration produces consistent electric fields and ECT dosing. Based on our results from the R61 investigation, individualized amplitude with right unilateral electrode placement has the potential to reliably achieve optimal dosing and will be tested with the R33 phase of the investigation.

Subjects will receive baseline imaging, clinical (primary outcome: clinician rated Inventory of Depressive Symptomatology, IDS-C30), and neuropsychological assessment (primary outcome: Delis Kaplan Executive Function System Verbal Fluency, DKEFS) 24 to 48 hours prior to the first ECT session (V1). Subjects will receive their second assessment (V2) one day after the sixth ECT treatment and the final assessment (V3) one day after the ECT series. If the subject fails to demonstrate improvement at V2 (< 25% reduction from baseline IDS-C30 total score, the primary antidepressant outcome), the subject will then receive bitemporal (BT) electrode placement for the remainder of the ECT series. The transition to BT will be a secondary antidepressant outcome. Subjects will be randomized to receive right unilateral (RUL) electrode placement with an individualized amplitude (n = 25) or traditional fixed 800 mA amplitude (n = 25, 1:1 ratio). Subjects and Raters will be blinded to subject assignment. Subjects in both arms will receive fixed pulse width (1.0 milliseconds), frequency (20 hertz), and pulse train duration (8 seconds).

For the individualized amplitude arm, subjects will receive RUL amplitude determined seizure titration during the first treatment like the R61 phase of the investigation (IDE for Soterix adapter: G200123). Subsequent RUL treatments will be completed with an individualized amplitude. To determine the individualized amplitude, we will use Ebrain. The individualized amplitude can be determined from the optimal E-field (V/m) / baseline E-field (V/m per mA). If a discrepancy exists between the amplitude seizure and E-field modeling methods that results in amplitude difference > 100 mA, we will use the E-field modeling method to determine the individualized amplitude. We will round the amplitude to the nearest 100 mA from 500 to 900 mA (the current dosing range of the FDA approved ECT device).

For the fixed 800 mA amplitude arm, subjects will receive RUL amplitude determined seizure titration during the first treatment. The rationale for amplitude titration with the fixed amplitude arm is to 1) improve the goodness of fit of the amplitude-seizure and Ebrain relationship; and 2) control for a sub-therapeutic stimulation associated with the first treatment for both arms. RUL amplitude seizure titration will be conducted during the first treatment like the individualized amplitude arm. Subsequent RUL treatments will be completed with 800 mA amplitude. The only difference between the arms will be individualized versus fixed 800 mA amplitude after amplitude titration.

A randomized controlled trial will compare hippocampal neuroplasticity, antidepressant, and cognitive outcomes between individualized amplitude and fixed 800 mA amplitude ECT in older depressed subjects (n = 25 per group, n = 50 total). Relative to fixed 800 mA ECT:

H1: Individualized amplitude arm will have improved RUL antidepressant outcome (IDS-C30 response rates and reduced BT electrode placement switch at V2).

H2: Individualized amplitude arm will have improved cognitive outcomes (DKEFS-Verbal Fluency

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder or bipolar II
* Clinical indications for ECT with right unilateral electrode placement

Exclusion Criteria:

* Defined neurological or neurodegenerative disorder (e.g., traumatic brain injury, epilepsy, Alzheimer's disease)
* Other psychiatric conditions (e.g., schizophrenia, bipolar I disorder)
* Current drug or alcohol use disorder (except for nicotine)
* Contraindications to MRI.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology - Clinician Rated | 4 weeks
  Depression severity, scores from 0 to 84, higher scores indicate more depression severity
Delis Kaplan Executive Function System Letter Fluency | 4 weeks
  Cognitive measure, scale scores range from 0 to 20, higher scores indicate better cognitive performance

CONTACTS AND LOCATIONS:
Overall Officials: Chris Abbott, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Science Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to National Data Archive.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after study completion.
Access Criteria: National Data Archive guidelines.